CLINICAL TRIAL: NCT00917800
Title: Diagnostic Benefits of HyperQ™ vs. Conventional ECG During Stress Test. A Comparison Study in Patients Referred for Angiography
Brief Title: Comparison of the HyperQ Versus Conventional Electrocardiogram (ECG) to Detect Ischemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: West German Heart Center Essen (Other)
Responsible Party: Principal Investigator, N. Reinsch, Principal Investigator, West German Heart Center Essen
Other Study IDs: Essen 09-3981
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Coronary Artery Disease
Keywords: angiography; exercise testing; high frequency ECG; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- suspected coronary artery disease: patients referred to angiography because of suspected coronary artery disease

SUMMARY:
The purpose of the investigation is to verify the efficiency of the HyperQ™ system in detecting exercise induced ischemia, with higher specificity and sensitivity than conventional ECG Stress testing. The study will be carried out by applying the HyperQ™ system during cycle ergometer stress testing in patients who are referred for angiography at the Department of Cardiology, Essen University Hospital, Essen, Germany. The HyperQ™ results will then be compared to the standard ECG stress test results using the angiography results as the gold standard. The study will be considered successful if analysis of the HyperQ provides a statistically significant improvement over the diagnostic accuracy of conventional ECG stress testing analysis.

ELIGIBILITY:
Inclusion Criteria:

* A patient who was referred to angiography.
* A patient who is able (i.e., no contraindications) to perform an exercise stress test
* A patient who signed an informed consent form.

Exclusion Criteria:

* Contraindications for an exercise test.
* Wolff-Parkinson-White (pre-excitation) syndrome.
* Left Bundle branch block, Complete Right bundle branch block or QRS duration > 120 ms, change in QRS morphology during exercise.
* Atrial Fibrillation or significant ventricular arrhythmia
* Treatment with Digoxin.
* Pacemaker.
* Having taken beta blockers within 24 hours before the exercise test.
* Pregnancy or suspected pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the West German Heart Center in Essen for coronary angiography
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the incremental diagnostic value of HyperQ data over exercise stress testing parameters to detect significant coronary artery disease (CAD) in patients referred for coronary angiography. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Erbel, MD, Principal Investigator — Director, West German Heart Center
Locations (1):
- West German Heart Center, Essen, Germany